CLINICAL TRIAL: NCT04213352
Title: Muscle Activation Of The Upper Trapezius During Computer Typing Task: A Comparison of Two Different Wrist Immobilization Methods
Brief Title: A Comparison of Two Different Wrist Immobilization Methods
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Halit SELÇUK, Research Assisstant, Marmara University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 31.10.2019/113
Record Dates: First submitted 2019-12-23; First posted 2019-12-30 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Work-Related Condition

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): The subjects will be asked to type on a computer for 5 minutes without splint or taping. The upper trapezius muscle activation will be recorded by surface EMG during the task. The mean values will be normalized according to Maximum Voluntary Isometric Contraction (MVIC) and %MVIC values.
- Splint Group (Experimental): The subjects will be asked to type on a computer for 5 minutes with a splint. The upper trapezius muscle activation will be recorded by surface EMG during the task. The mean values will be normalized according to Maximum Voluntary Isometric Contraction (MVIC) and %MVIC values.
  Interventions: Other: Wrist Splint
- Rigid Taping Group (Experimental): The subjects will be asked to type on a computer for 5 minutes with rigid taping which limits the wrist flexion at the dominant side. The upper trapezius muscle activation will be recorded by surface EMG during the task. The mean values will be normalized according to Maximum Voluntary Isometric Contraction (MVIC) and %MVIC values.
  Interventions: Other: Rigid Taping

INTERVENTIONS:
Other: Wrist Splint — Neutral position and volar supported wrist orthosis which limits the flexion and deviation while allowing pronation, supination, and extension of the wrist.
  Arms: Splint Group
Other: Rigid Taping — Rigid taping in the neutral position will be performed to allow pronation, supination, and extension of the wrist while limiting the flexion and deviation.
  Arms: Rigid Taping Group

SUMMARY:
The aim of this study is to examine the effect of the splint and rigid taping on the muscle activation of the upper trapezius muscle during computer typing tasks in office workers.

The study will be conducted on 10 healthy office workers. The study subjects will be asked to type on a computer for 5 minutes (1) without splint or taping, (2) with a splint and (3) with rigid taping which limits the wrist flexion at the dominant side. The upper trapezius muscle activation will be recorded by surface EMG during the task. The mean values will be normalized according to Maximum Voluntary Isometric Contraction (MVIC) and %MVIC values.

ELIGIBILITY:
Inclusion Criteria:

* Being an office worker between 20-35 years of age
* Using a computer for at least 4 hours a day
* Working full time for at least 1 year without any upper extremity pathology

Exclusion Criteria:

* Having a body mass index of 30 kg / m2 or more on the day of evaluation
* Using muscle relaxants 72 hours before the evaluation
* Exercising within the last 48 hours

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-01-10 (Estimated); Primary Completion 2020-02-01 (Estimated); Study Completion 2020-02-15 (Estimated)

PRIMARY OUTCOMES:
Measurement of Muscle Activation for Control Group | It will be recorded at baseline for MVIC and 1 minute after baseline while performing the 5-minute typing task on computer for %MVIC
  Surface Electromyography (sEMG) device will be used for measurement of muscle activation. The electrodes going to be placed according to the SENIAM criteria(1). First, the MVIC will be performed by each individual in the manual muscle testing position. 6 seconds MVIC will be measured with 3 repetitions and a 3-minute rest period going to be given. The highest value of the three measurements will be recorded as MVIC. The computer task consists of typing 300-word text for 5 minutes. Individuals will be instructed about the typing task and to be seated comfortably and as close to screen as possible. The 5-minute typing task will be performed without orthosis or taping. The upper trapezius muscle activation will be recorded with the sEMG. The number of words participants wrote will be noted. To prevent muscle fatigue, a resting period of 5 minutes will be given. The mean values (mV) during the writing task with sEMG will be normalized according to MVIC and %MVIC values will be determined.
Measurement of Muscle Activation for Splint Group | It will be recorded at baseline for MVIC and 1 minute after baseline while performing the 5-minute typing task on computer for %MVIC
  Surface Electromyography (sEMG) device will be used for measurement of muscle activation. The electrodes going to be placed according to the SENIAM criteria(1). First, the MVIC will be performed by each individual in the manual muscle testing position. 6 seconds MVIC will be measured with 3 repetitions and a 3-minute rest period going to be given. The highest value of the three measurements will be recorded as MVIC. The computer task consists of typing 300-word text for 5 minutes. Individuals will be instructed about the typing task and to be seated comfortably and as close to screen as possible. The 5-minute typing task will be performed with orthosis. The upper trapezius muscle activation will be recorded with the sEMG. The number of words participants wrote will be noted. To prevent muscle fatigue, a resting period of 5 minutes will be given. The mean values (mV) during the writing task with sEMG will be normalized according to MVIC and %MVIC values will be determined.
Measurement of Muscle Activation for Rigid Taping Group | It will be recorded at baseline for MVIC and 10 minutes after baseline while performing the 5-minute typing task on computer for %MVIC
  Surface Electromyography (sEMG) device will be used for measurement of muscle activation. The electrodes going to be placed according to the SENIAM criteria(1). First, the MVIC will be performed by each individual in the manual muscle testing position. 6 seconds MVIC will be measured with 3 repetitions and a 3-minute rest period going to be given. The highest value of the three measurements will be recorded as MVIC. The computer task consists of typing 300-word text for 5 minutes. Individuals will be instructed about the typing task and to be seated comfortably and as close to screen as possible. The 5-minute typing task will be performed with rigid taping. The upper trapezius muscle activation will be recorded with the sEMG. The number of words participants wrote will be noted. To prevent muscle fatigue, a resting period of 5 minutes will be given. The mean values (mV) during the writing task with sEMG will be normalized according to MVIC and %MVIC values will be determined.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hermens HJ, Freriks B, Disselhorst-Klug C, Rau G. Development of recommendations for SEMG sensors and sensor placement procedures. J Electromyogr Kinesiol. 2000 Oct;10(5):361-74. doi: 10.1016/s1050-6411(00)00027-4. PMID 11018445